CLINICAL TRIAL: NCT07015788
Title: Open -Label,Cross Over Trail Evaluating the Glycemic Impact of Peach Varieties in Healthy Adullts
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rehman Medical Institute - RMI (Other)
Responsible Party: Principal Investigator, Naseer Ahmed, Associate proffesor, Rehman Medical Institute - RMI
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GL/GI-NA_1V5
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-05

CONDITIONS: Blood Glucoe
Keywords: glycemic index; glycemic load
MeSH Terms: interventions — CD44 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group (cross over) (Active Comparator): Participants will consume 50 grams of glucose solution. This serves as the reference standard for calculating glycemic index values of the peach varieties.
  Interventions: Other: EARLY GRAND; Other: SPRING CREST PEACH; Other: INDIAN BLOOD

INTERVENTIONS:
Other: EARLY GRAND — Participants will consume a standardized portion of peach variety A containing 50 grams of available carbohydrates. Capillary blood glucose levels will be measured at multiple time points post-consumption to assess glycemic response.
Other: SPRING CREST PEACH — Participants will consume a standardized portion of peach variety B containing 50 grams of available carbohydrates. Capillary blood glucose levels will be measured at multiple time points post-consumption to assess glycemic response.
Other: INDIAN BLOOD — Participants will consume a standardized portion of peach variety C containing 50 grams of available carbohydrates. Capillary blood glucose levels will be measured at multiple time points post-consumption to assess glycemic response.

SUMMARY:
This study aims to evaluate the effect of different peach varieties on the glycemic index (GI) in healthy adult participants. While peaches are generally classified as low-GI fruits, variations in sugar composition, fiber content, and ripeness among different cultivars may influence their glycemic response. By assessing and comparing the GI values of several commonly consumed peach varieties, this trial seeks to provide more precise dietary recommendations for glycemic control and support better fruit selection for individuals managing blood glucose levels.

DETAILED DESCRIPTION:
This study aims to evaluate the effect of different peach varieties on the glycemic index (GI) in healthy adult participants. While peaches are generally classified as low-GI fruits, variations in sugar composition, fiber content, and ripeness among different cultivars may influence their glycemic response. By assessing and comparing the GI values of several commonly consumed peach varieties, this trial seeks to provide more precise dietary recommendations for glycemic control and support better fruit selection for individuals managing blood glucose levels.

ELIGIBILITY:
Inclusion Criteria:• Healthy male and female adults aged 18-50 years

* BMI between 18.5-24.9 kg/m²
* Normal fasting blood glucose (<100 mg/dL)
* Willingness to adhere to the study protocol Exclusion Criteria:• Diagnosed diabetes, metabolic syndrome, or any glucose metabolism disorder
* Use of medications or supplements that affect glucose levels
* Allergy to peaches or intolerance to test/reference foods
* Pregnant or breastfeeding women
* Smoking or use of recreational drugs

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Glycemic Index | 2 hours post-consumption (per intervention)
  Participants will consume a standardized portion of a peach variety containing 50 grams of available carbohydrates. Capillary blood glucose levels will be measured at multiple time points post-consumption to assess glycemic response.

SECONDARY OUTCOMES:
Incremental Area Under the Curve (iAUC) for Blood Glucose | 0-120 minutes post-consumption
  The iAUC will be calculated for each intervention using the trapezoidal method, excluding values below baseline. This helps quantify the glycemic response.
Peak Blood Glucose Concentration | 0-120 minutes post-consumption
  The highest recorded blood glucose concentration during the 2-hour postprandial period following consumption of each intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Rehman Medical Institue, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Basit et al. (2022). J Pak Med Assoc. (Health burden).
- [Background] IDF Diabetes Atlas 2021 (Pakistan ranked 3rd in diabetes cases).